CLINICAL TRIAL: NCT02805868
Title: A Single-arm, Single Center, Pilot Study of Siltuximab, an Anti-IL6 Therapy, for Patients With Myelofibrosis
Brief Title: Siltuximab in Treating Patients With Primary, Post-Polycythemia Vera, or Post-Essential Thrombocythemia Myelofibrosis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16H01; STU00202680 (CTRP (Clinical Trial Reporting Program)); NU 16H01 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00685 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Myelofibrosis; Polycythemia Vera; Primary Myelofibrosis; Thrombocytopenia
Keywords: Severe; Anemia; Aplastic; Post-Polycythemic; Transformation; Thrombocythemia; Essential
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocytopenia; Lymphoma, Follicular; Anemia; Thrombocytosis | interventions — Biopsy; siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (siltuximab) (Experimental): Patients receive siltuximab IV over 60 minutes on day 1. Patients also undergo bone marrow biopsy and aspiration at baseline and at the end of treatment (within 30 days of last siltuximab dose) or as clinically indicated. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who are responding after 6 courses may receive additional siltuximab treatment for up to 1 year at the discretion of the study doctor.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Other: Laboratory Biomarker Analysis; Biological: Siltuximab

INTERVENTIONS:
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Siltuximab — Given IV
  Other Names: Anti-IL-6 Chimeric Monoclonal Antibody; cCLB8; CNTO 328; CNTO-328; Sylvant

SUMMARY:
The main purpose of this investigational research study is to determine how safe and tolerable the study drug siltuximab is in patients with myelofibrosis (MF). This medication has been approved by the FDA for another condition (multicentric castleman's disease (MCD), but not for myelofibrosis (MF). In MCD, siltuximab resulted in improvement in symptoms and anemia. While MCD and MF are different diseases, they share some common features including a protein call interleukin-6 (IL-6) that may be important in causing symptoms of MCD and MF.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety and tolerability of the drug siltuximab in the myelofibrosis patient population.

SECONDARY OBJECTIVES:

I. To determine clinical improvement (CI). II. To determine the overall response rate (ORR).

TERTIARY OBJECTIVES:

I. To determine if siltuximab results in improvement in iron dysregulation. II. To determine changes in inflammatory stress that may correlate with clinical response.

OUTLINE:

Patients receive siltuximab intravenously (IV) over 60 minutes on day 1. Patients also undergo bone marrow biopsy and aspiration at baseline and at the end of treatment (within 30 days of last siltuximab dose) or as clinically indicated. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression, unacceptable toxicity, or patient decision to withdraw. Patients who are responding after 6 courses may receive additional siltuximab treatment for up to 1 year at the discretion of the study doctor.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of primary myelofibrosis (PMF), post-polycythemia vera (post-PV) myelofibrosis (MF), or post-essential thrombocythemia (post-ET) MF using World Health Organization Criteria
* Patients must have disease that requires therapy, including intermediate-1, intermediate-2, or high-risk disease according to the International Prognostic Scoring System (IPSS) or Dynamic-IPSS
* Patients must be off myeloproliferative neoplasm (MPN) directed therapy, such as Janus kinase (JAK)-inhibitors, for at least 2 weeks prior to administration of the study drug; NOTE: This does not include supportive transfusion, or hydroxyurea; these must be stopped prior to first day of treatment, but no wash -out period is required
* Patients must be resistant to, intolerant of, or ineligible for JAK2 inhibitor therapy, based on severe anemia or thrombocytopenia
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* New York Heart Association functional classification for congestive heart failure (NYHA CHF) < 3
* Patients must have clinical laboratory values meeting the following criteria within 28 days prior to registration:
* Absolute neutrophil count >= 1.0 x 10^9/L (without growth factor support)
* Platelet count >= 20 x 10^9/L (without transfusion support within 2 weeks of registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 x ULN
* Total bilirubin =< 2.5 x upper limit of normal (ULN) except if the elevation is due to Gilbert's syndrome (allowable at =< 5 x ULN) or myelofibrosis (per principle investigator [PI] discretion)
* Calculated creatinine clearance > 20 mL/min per institutional standard
* Before enrollment, a woman must be one of the following:

  * Not of childbearing potential, defined as:

    * Postmenopausal (> 45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level > 40 IU/mL)
    * Permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy)
    * Otherwise be incapable of pregnancy
  * Of childbearing potential and practicing a highly effective method of birth control (consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies) during the study and for 3 months after receiving the last dose of study agent NOTE: Examples include established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidals (including foam/gel/film/cream/suppository) or occlusive cap (diaphragm or cervical/vault caps) with spermicidals; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject); Note: If the childbearing potential changes after start of the study (e.g., woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above
* Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to registration
* Female patients must agree (during the study and for 3 months after receiving the last dose of study agent, not to donate eggs (ova, oocytes) for the purposes of assisted reproduction
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidals or partner with occlusive cap with spermicidals and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Patients with prior exposure to agents targeting interleukin 6 (IL -6) or the IL-6 receptor are not eligible
* Patients with another malignancy, unless they have been disease free for 2 years prior to registration, with the exception of

  * Basal cell or non-metastatic squamous cell carcinoma of the skin
  * Cervical carcinoma in situ or International Federation of Gynecology and Obstetrics (FIGO) stage 1 carcinoma of the cervix
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring concurrent systemic antibiotic treatment: there is no mandatory duration of time that a patient has to be off antibiotics, but the treating physician has to deem the infection as effectively treated prior to enrollment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients who have received vaccination with live attenuated vaccines within 6 months prior to registration are not eligible
* Patients who are on any prohibited medication; they have to be have a wash-out period of at least 2 weeks prior to registration, in order to be eligible for the study
* Patients with clinically significant infection, including known human immunodeficiency virus (HIV), human herpesvirus-8 (HHV-8), hepatitis C infection, or known hepatitis B surface antigen positivity are not eligible
* Female patients who are pregnant or breast-feeding are not eligible; NOTE: A woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study agent should likewise not be considered for this study
* Patients who have received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half -lives before registration or is currently enrolled in the treatment stage of an investigational study are not eligible; please contact PI for further details on wash-out period and eligibility of such patients
* Patients who have been hospitalized for infection or major surgery (e.g., requiring general anesthesia) within 2 weeks before registration or have not fully recovered from surgery are not eligible; Note: Subjects with surgical procedures conducted under local anesthesia may participate
* Patients who are unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 30 days after last treatment
  To evaluate safety and tolerability of the drug siltuximab in the myelofibrosis patient population. Adverse events will be assessed by type, timing, frequency, and attribution and will be graded according to the NCI's common terminology criteria, version 4.03.

SECONDARY OUTCOMES:
Clinical Improvement (CI): changes in symptoms | At baseline and after cycle 3 (9 weeks)
  Changes in the baseline symptom burden using Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) questionnaire.
Clinical Improvement (CI): splenomegaly | At baseline and after cycle 3 (9 weeks)
  To determine spleen response, palpation will be used, using centimeters below the left costal margin, and if body habitus is prohibitive, by ultrasonography.
Clinical Improvement (CI): Anemia response | At baseline and after cycle 3 (9 weeks)
  Baseline hemoglobin level and/or transfusion-dependence will be recorded at baseline and compared to results after cycle 3
Overall Response Rate (ORR) | After 6 cycles of treatment (18 weeks)
  The ORR will be assessed after 6 cycles of therapy using standard criteria published by the International Working Group for Myelofibrosis Research and Treatment which will evaluate for complete response, partial response, clinical improvement, or stable disease.

OTHER OUTCOMES:
Iron Dysregulation | At baseline, after cycle 3 (9 weeks), and after cycle 6 (18 weeks)
  Peripheral blood will be taken to determine if siltuximab results in improvement in iron dysregulation.
Changes in inflammatory stress: C-reactive protein (CRP) | At baseline, after cycle 3 (9 weeks), and after cycle 6 (18 weeks)
  To determine changes in inflammatory stress that may correlate with clinical response. To assess this, CRP will be measured.
Changes in inflammatory stress: hepcidin levels | At baseline, after cycle 3 (9 weeks), and after cycle 6 (18 weeks)
  To determine changes in inflammatory stress that may correlate with clinical response. To assess this, hepcidin will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Brady Stein, MD, Principal Investigator — Northwestern University